CLINICAL TRIAL: NCT02728700
Title: Pilot Safety and Feasibility Trial of Mycophenolate and Sirolimus for Prevention of GVHD in Mismatched Unrelated and Related Donor Hematopoietic Stem Cell Transplantation for Hematologic Malignancies
Brief Title: Sirolimus and Mycophenolate Mofetil in Preventing GVHD in Patients With Hematologic Malignancies Undergoing HSCT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual factor
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-34973; NCI-2016-00387 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEDSBMT295 (Other: OnCore)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Adult Hodgkin Lymphoma; Adult Myelodysplastic Syndrome; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Childhood Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Childhood Hodgkin Lymphoma; Childhood Myelodysplastic Syndrome; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Myelofibrosis; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Non-Hodgkin Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Non-Hodgkin Lymphoma; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Anemia, Refractory, with Excess of Blasts; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (sirolimus, HSCT, MMF) (Experimental): Patients receive sirolimus PO starting on day -3, 3 times a week during hospitalization and then once a week for up to 6 months. Patients undergo HSCT on day 0. Patients also receive mycophenolate mofetil IV or PO TID on days 1-180. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Drug: Sirolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given IV
  Other Names: Cellcept; MMF
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; RAPAMYCIN; SILA 9268A; WY-090217

SUMMARY:
This pilot phase I/II trial studies the side effects and how well sirolimus and mycophenolate mofetil work in preventing graft versus host disease (GvHD) in patients with hematologic malignancies undergoing hematopoietic stem cell transplant (HSCT). Biological therapies, such as sirolimus and mycophenolate mofetil, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop tumor cells from growing. Giving sirolimus and mycophenolate mofetil after hematopoietic stem cell transplant may be better in preventing graft-versus-host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and feasibility of administering sirolimus and mycophenolate mofetil (MMF) as prophylaxis of grade III-IV acute graft versus host disease (aGvHD) in patients undergoing mismatched unrelated and related donor hematopoietic stem cell transplant (HSCT).

OUTLINE:

Patients receive sirolimus orally (PO) starting on day -3, 3 times a week during hospitalization and then once a week for up to 6 months. Patients undergo HSCT on day 0. Patients also receive mycophenolate mofetil intravenously (IV) or PO three times a day (TID) on days 1-180. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at days 30, 60, 100, 180, 270, and 365, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have one of the following disease categories:

  * Acute myeloid leukemia (AML) beyond 2nd remission or relapsed/refractory disease
  * Acute lymphoblastic leukemia (ALL) beyond 2nd remission or relapsed/refractory disease
  * Chronic myeloid leukemia (CML) beyond 2nd chronic phase or in blast crises
  * Myelodysplastic syndrome (MDS)
  * Myeloproliferative disorders including myeloid metaplasia and myelofibrosis
  * High risk non-Hodgkin's lymphoma (NHL) in first remission
  * Relapsed or refractory NHL
  * Hodgkin's lymphoma (HL) beyond first remission
* Performance status by Karnofsky of >= 70% or Lansky > 70% for patients < 16 years of age
* Human leukocyte antigen (HLA) mismatched related or unrelated donor identified 8/10 or 9/10
* Willingness to take oral medications during the transplantation period
* Willingness and ability to sign a written informed consent (assent if applicable)

Exclusion Criteria:

* Prior myeloablative allogeneic or autologous HSCT
* Human immunodeficiency virus (HIV) infection
* Pregnant or lactating females
* Evidence of uncontrolled active infection
* Down syndrome
* Serum creatinine (CR) < 1.5mg/dl or 24 hour CR clearance < 50 ml/min
* Direct bilirubin > 2 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x ULN
* Carbon monoxide diffusing capability test (DLCO) > 60% predicted and in children- room air oxygen saturation > 92%
* Left ventricular ejection fraction < 45% and in children-shortening fraction < 26%
* Fasting cholesterol > 300 mg/dl or triglycerides > 300 while on lipid lowering agents
* Patients who have received an investigational drug within 30 days of enrollment in study
* Patients with prior malignancies except basal cell carcinoma or treated carcinoma in-situ; cancer treated with curative intent > 5 years will be allowed; cancer treatment with curative intent =< 5 years will not be allowed

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GvHD grade 3 & 4, according to the Glucksberg staging criteria | Up to 60 days post-transplant
  Statistical analysis results will be reported using summary tables, figures, and data listings. Continuous variables will be summarized using the mean, standard deviation, median, minimum, and maximum.
Incidence of acute GvHD grade 3 & 4, according to the Glucksberg staging criteria | Up to 100 days post-transplant
  Statistical analysis results will be reported using summary tables, figures, and data listings. Continuous variables will be summarized using the mean, standard deviation, median, minimum, and maximum.

SECONDARY OUTCOMES:
Incidence of thrombotic microangiopathy defined according to the bone marrow transplant clinical trials network toxicity committee | Up to 100 days
  Defined as: red blood cell fragmentation and at least two schistocytes per high-power field on peripheral smear; concurrent increased serum lactate dehydrogenase measurement above institutional baseline; concurrent doubling of serum creatinine or 50% increase in creatinine clearance from baseline and/or neurological dysfunction without other explanations; and negative direct and indirect Coombs. Statistical analysis results will be reported using summary tables, figures, and data listings. Continuous variables will be summarized using the mean, standard deviation, median, minimum, and maximum.
Incidence of venous-occlusive disease (VOD) using Modified Seattle Criteria | Up to 100 days
  Severe VOD will be considered a dose limiting toxicity. Statistical analysis results will be reported using summary tables, figures, and data listings. Continuous variables will be summarized using the mean, standard deviation, median, minimum, and maximum.
Severity of mucositis determined by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 100 days
  Grade III and IV will be considered dose limiting toxicities. Statistical analysis results will be reported using summary tables, figures, and data listings. Categorical variables will be summarized by numbers and percentages of subjects in corresponding categories.
Time to neutrophil engraftment defined as first of 3 consecutive days with the absolute neutrophil count is > 500/ul in the peripheral blood | Baseline to up to 100 days
  Statistical analysis results will be reported using summary tables, figures, and data listings. Continuous variables will be summarized using the mean, standard deviation, median, minimum, and maximum.
Time to platelet engraftment defined as the first day of a minimum of three consecutive measurements on different days when platelet count > 50,000/mm^3 and patient is transfusion-independent for a minimum of 7 days | Baseline to up to 100 days
  Statistical analysis results will be reported using summary tables, figures, and data listings. Continuous variables will be summarized using the mean, standard deviation, median, minimum, and maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Agarwal-Hashmi, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No